CLINICAL TRIAL: NCT02210676
Title: Residual Extensor Lag Approximately 1 Month After Splint or Cast Immobilization of a Mallet Finger
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the investigator leaving the institution, the study was terminated
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David C. Ring, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014P001041
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Patients Present With Mallet Finger

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with Mallet Finger (Experimental): All enrolled patients
  Interventions: Other: PROMIS Upper Extremity; Other: Likert Pain Scale; Other: Mallet Finger Extensor Lag Measurement

INTERVENTIONS:
Other: PROMIS Upper Extremity
Other: Likert Pain Scale
Other: Mallet Finger Extensor Lag Measurement

SUMMARY:
Aim:

The purpose of the study is to learn more about how a person recovers after treatment for mallet finger injury. The investigators want to identify the best outcome after mallet finger injury and how to improve treatment strategies.

Primary null hypothesis:

There are no statistically significant factors associated with extensor lag between 4 weeks and 4 months after immobilization is discontinued for a mallet finger among demographic, injury, and treatment factors.

Secondary null hypothesis:

There are no statistically significant factors associated with PROMIS upper extremity function between 4 weeks and 4 months after completion of immobilization for a mallet finger among demographic, psychological, injury, and treatment factors.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* English fluency and literacy
* Mallet finger fracture or non-fracture
* Mallet finger subluxation or non-subluxation

Exclusion Criteria:

* Pregnant Women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Mallet Finger Extensor Lag | Baseline
Mallet Finger Extensor Lag | 4 weeks to 4 months after diagnosis

SECONDARY OUTCOMES:
Patient Reported Outcomes Measure Information System (PROMIS) Upper Extremity | 4 weeks to 4 months after diagnosis
  A computerized assessment of upper extremity function
Likert Pain Scale | 4 weeks to 4 months after diagnosis
Demographics Questionnaire | 4 weeks to 4 months after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States